CLINICAL TRIAL: NCT01473810
Title: Immunotherapy of HIV-infected Patients: A Single-blinded, Randomized, Immunogenicity, Pilot Study of Intranasal Administration of Vacc-4x With Endocine as Adjuvant
Brief Title: Intranasal Modified Vacc-4x Gag Peptides With Endocine as Adjuvant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Bionor Immuno AS (Industry); Eurocine Vaccines AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CTN-Vacc-4x/L3-2011/1
Record Dates: First submitted 2011-11-01; First posted 2011-11-17 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: HIV Infection
Keywords: HIV; vaccination; T cells; mucosal immunity; safety; nasal administration; DTH skin test
MeSH Terms: conditions — HIV Infections | interventions — Vacc-4x; Endocine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vacc-4x low dose (Experimental): 80 µg Vacc-4x (20 µg pr. peptide) in 300 µl Endocine divided into two administrations, one for each nose cavity
  Interventions: Biological: Vacc-4x low dose
- Vacc-4x medium dose (Experimental): 400 µg Vacc-4x (100 µg pr. peptide) in 300 µl Endocine divided into two administrations, one for each nose cavity
  Interventions: Biological: Vacc-4x medium dose
- Vacc-4x high dose (Experimental): 1200 µg Vacc-4x (300 µg pr. peptide) in 300 µl Endocine divided into two administrations, one for each nose cavity
  Interventions: Biological: Vacc-4x high dose
- Zero dose (Placebo Comparator): Adjuvant only, i.e. 300 µl Endocine divided into two administrations, one for each nose cavity
  Interventions: Biological: Zero dose

INTERVENTIONS:
Biological: Vacc-4x low dose — 80 µg Vacc-4x (20 µg pr. peptide) in 300 µl Endocine divided into two administrations, one for each nose cavity, administrated once weekly for four weeks
  Other Names: Vacc-4x; Endocine
  Arms: Vacc-4x low dose
Biological: Vacc-4x medium dose — 400 µg Vacc-4x (100 µg pr. peptide) in 300 µl Endocine divided into two administrations, one for each nose cavity, administrated once weekly for four weeks
  Other Names: Vacc-4x; Endocine
  Arms: Vacc-4x medium dose
Biological: Vacc-4x high dose — 1200 µg Vacc-4x (300 µg pr. peptide) in 300 µl Endocine divided into two administrations, one for each nose cavity, administrated once weekly for four weeks
  Other Names: Vacc-4x; Endocine
  Arms: Vacc-4x high dose
Biological: Zero dose — 300 µl Endocine divided into two administrations, one for each nose cavity, administrated once weekly for four weeks
  Other Names: Endocine
  Arms: Zero dose

SUMMARY:
HIV-specific cellular immunity is hampered in most HIV-infected individuals. Therapeutic immunization in HIV aims to strengthen the HIV-specific cellular immunity, usually in the absence of replicating HIV with antiretroviral drugs. The aims of this strategy can be to decrease the mass of latently infected CD4+ T cells, better tolerance of drug-free periods, and better select candidates for preventive HIV vaccines.

Vacc-4x is one of the few peptide-based therapeutic vaccines tested, and consists of four, slightly modified HIV Gag p24 consensus peptides. Vacc-4x was first tested by intradermal injections using GM-CSF as adjuvant. A recent multinational placebo-controlled study found improvement of vaccine-specific T cell immunity and decrease in viral loads (presented at the AIDS vaccine 2011 conference, Bangkok).

In this study the investigators hypothesize that the Vacc-4x peptides, deposited on the nasal mucosal surfaces in conjunction with Endocine, a newly developed and documented mucosal adjuvant, will induce T cell responses to HIV and improve HIV-specific immunity both systemically and at mucosal surfaces (oral, rectal, vaginal).

DETAILED DESCRIPTION:
HIV-specific cellular immunity is hampered in most HIV-infected individuals, partly because the virus infects CD4+ T cells, the key cell subset in all immune responses. CD4 is the primary HIV receptor (CD4), but infection requires a co-receptor (CCR5) which is carried mainly by activated T cells. During primary HIV-infection, two types of CD4+ T cells mainly become infected: (i) Sub-activated T cells of all specificities within the mucosal linings, particularly in the gut; and (ii) HIV-specific T cell clones, that proliferates and are activated as a normal response to HIV infection itself. The HIV-specific immunity therefore becomes severely compromised early in the infection. Patients having better T cells specific to parts of the HIV Gag matrix protein usually progress slower towards AIDS than patients with poor T cell responsitivity towards Gag.

Therapeutic immunization in HIV aims to strengthen the HIV-specific cellular immunity, usually in the absence of replicating HIV with antiretroviral drugs. The aims of this strategy can be to decrease the mass of latently infected CD4+ T cells, better tolerance of drug-free periods, and better select candidates for preventive HIV vaccines. The latter point may be important since clinical trials with preventive vaccine candidates may challenge our ethical standards: Such trials must be very large and conducted in poor areas with high prevalence of HIV, in order to have as many (placebo) or few (vaccine candidate) new HIV infections as fast as possible. Preventive vaccine trials might therefore compete with introduction of "western" access to HIV drugs.

Vacc-4x is one of the few peptide-based therapeutic vaccines tested, and consists of four, slightly modified HIV Gag p24 consensus peptides. Vacc-4x was first tested by intradermal injections using GM-CSF as adjuvant. In a dose study at our Hospital, the investigators found induction of robust cellular immune responses both in vitro and in vivo by skin testing, indications of improved viral control, long-lasting immunity and lack of mutational changes in the HIV strains within the study cohort. A recently completed multinational placebo-controlled study found improvement of viral loads (presented at the AIDS vaccine 2011 conference, Bangkok).

In this study the investigators hypothesize that the Vacc-4x peptides, deposited on the nasal mucosal surfaces in conjunction with Endocine, a newly developed and documented mucosal adjuvant, will induce T cell responses to HIV and improve HIV-specific immunity both systemically and at mucosal surfaces (oral, rectal, vaginal). This route of application may even simplify mass vaccination. The study is primarily a dose-study focused on adverse events, which have been negligible when Vacc-4x was given parenterally, as well as induction of systemic and mucosal immunity.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years, both genders.
* HIV positive at least one year.
* Clinically stable on ART for the last 6 months (changes in therapy is allowed as long as the viral load is stable).
* Documented viral load (HIV-1 RNA) less than 50 copies/mL for the last six months.
* Documented stable CD4 cell count ≥ 400x106/L.
* Nadir (lowest ever) CD4 cell count ≥ 200x106/L.
* Signed informed consent.

Exclusion Criteria:

* Reported pre-study AIDS-defining illness within the previous year.
* Malignant disease.
* On chronic treatment with immunosuppressive therapy.
* Unacceptable values of the hematologic and clinical chemistry parameters, as judged by the Principle Investigator (or designee), including creatinine values >1.5x upper limit of normal (ULN), and AST (SGOT), ALT (SGPT) and alkaline phosphatase values >2.5x ULN.
* Concurrent chronic active infection such as chronic viral hepatitis B or C or active tuberculosis.
* Pregnant or breastfeeding women.
* Women of childbearing potential not using reliable and adequate contraceptive methods (defined as: use of oral, implanted, injectable, mechanical or barrier products for the prevention of pregnancy; practicing abstinence; sterile) during the study, or sexually active male patients with partners of childbearing potential unwilling to practice effective contraception during the study.
* Current participation in other clinical therapeutic studies.
* Incapability of compliance to the treatment protocol, in the opinion of the Investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of intranasal administration of Vacc-4x with Endocine as adjuvant at three different dose levels | 2 months after completion of last patient.
  Record adverse events including severe adverse events according to GCP

SECONDARY OUTCOMES:
Evaluate cellular immune response to Vacc-4x in vivo by Vacc-4x DTH skin test | Up to 2 months after completion of last patient
  Record intradermal Vacc-4x-associated delayed-type hypersensitivity test (DTH) in vivo by measuring skin induration (area) 2 days after injecion qt end of study week 8, in comparison with 38 historical unvaccinated HIV seropositive controls
Evaluate cellular immune response to Vacc-4x in vitro | Up to 6 months after completion of last patient
  Measure changes in Vacc-4x-specific T cell proliferation and activation compared with baseline values for each individual participant, i.e. before vaccination
Evaluate the effect on CD4+ T cell counts and viral load (HIV-1 RNA) in peripheral blood | Up to 2 months after completion of last patient
  Measure individual changes in CD4 counts and viral loads at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dag Kvale, Professor/MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Department of Infectious Diseases, Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Brekke K, Lind A, Holm-Hansen C, Haugen IL, Sorensen B, Sommerfelt M, Kvale D. Intranasal administration of a therapeutic HIV vaccine (Vacc-4x) induces dose-dependent systemic and mucosal immune responses in a randomized controlled trial. PLoS One. 2014 Nov 14;9(11):e112556. doi: 10.1371/journal.pone.0112556. eCollection 2014. PMID 25398137
- See also: University of Oslo, Faculty of Medicine, public web page for PI — http://www.med.uio.no/klinmed/personer/vit/dagkv/index.html
- See also: Web page of Vacc-4x vaccine patent holder (not sponsor, peptide supply free of charge, research collaborator) — http://www.bionorimmuno.com/
- See also: Web page of adjuvant patent holder (not sponsor, research collaborator, expenses in part covered by Research Council of Norway) — http://www.eurocine-vaccines.com/